CLINICAL TRIAL: NCT01872052
Title: Dipole Density Right Atrial Mapping and Assessment of Therapy In Cavotricuspid Isthmus Flutter
Acronym: DDRAMATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CL-AFL-001
Record Dates: First submitted 2013-05-02; First posted 2013-06-07 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Acutus Medical System (Experimental)
  Interventions: Device: Acutus Medical System Mapping

INTERVENTIONS:
Device: Acutus Medical System Mapping — Mapping with the Acutus Medical System followed by intracardiac ablation of typical atrial flutter

SUMMARY:
Study to determine the feasibility of the Acutus Medical System in obtaining data to create Dipole Density Maps of electrical activation in the right atrium in patients with typical atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* One documented occurrence of typical AFL within the past 6 months
* Be able and willing to sign informed consent

Exclusion Criteria:

* Contraindication to a non-emergent interventional EP procedure
* Require treatment in or access to left atrium
* Had a myocardial infarction within the prior two months
* Had cardiac surgery within the prior three months
* Intracardiac thrombus
* Permanent pacemaker/ICD leads in/through right atrium
* Clinically significant tricuspid valve regurgitation or stenosis
* Cerebral ischemic event (including TIA) in the prior six months
* Pregnant
* Currently enrolled in any other clinical investigation
* Any other significant uncontrolled or unstable medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The number of patients in which offline construction of pre- and post-treatment activation maps can be completed | 3 months post-procedure
  Proprietary software algorithms will be used generate electrical activation maps based dipole density data acquired by the Acutus Medical Catheter during the procedures. These activation maps will then be applied to a 3D model of the endocardial surface to create a 3D activation map.
The number of patients that experience a device-related adverse events as a measure of safety and tolerability | 7 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- AZ Sint-Jan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: Undecided